CLINICAL TRIAL: NCT01229761
Title: A Randomized Study of Cotrimoxazole Prophylaxis and Longer Breastfeeding Duration to Improve Survival Among HIV-Exposed Infants in Botswana
Brief Title: Study to Improve Survival Among HIV-Exposed Infants in Botswana
Acronym: Mpepu
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Roger Shapiro, Principal Investigator, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 18677; R01HD061265 (NIH)
Record Dates: First submitted 2010-10-22; First posted 2010-10-28 (Estimated); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: HIV Infections; Neutropenia; Anemia
Keywords: HIV; Trimethoprim-Sulfamethoxazole Combination; Breast Feeding; Infant Mortality; Morbidity; Botswana; Africa; Infectious disease transmission, vertical; adverse drug event
MeSH Terms: conditions — HIV Infections; Neutropenia; Anemia; Breast Feeding; Infant Death; Drug-Related Side Effects and Adverse Reactions | interventions — Trimethoprim, Sulfamethoxazole Drug Combination; Aging; Lactation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- infant cotrimoxazole (Active Comparator)
  Interventions: Drug: cotrimoxazole prophylaxis
- infant placebo (Placebo Comparator)
  Interventions: Drug: cotrimoxazole placebo
- exclusive breastfeeding for 6 months (Active Comparator)
  Interventions: Behavioral: exclusive breastfeeding until 6 months of age
- exclusive breastfeeding for 12 months (Active Comparator)
  Interventions: Behavioral: breastfeeding for 12 months

INTERVENTIONS:
Drug: cotrimoxazole prophylaxis — 100mg/20mg per day (or 2.5 mL of syrup from a 200mg/40mg per 5mL suspension) from 1-6 months, followed by 200mg/40mg per day (or 5 mL of syrup from a 200mg/40mg per 5 mL suspension) from 6 to 12 months
  Other Names: Trimethoprim-Sulfamethoxazole Combination
  Arms: infant cotrimoxazole
Drug: cotrimoxazole placebo — 100mg/20mg per day (or 2.5 mL of syrup from a 200mg/40mg per 5mL suspension) from 1-6 months, followed by 200mg/40mg per day (or 5 mL of syrup from a 200mg/40mg per 5 mL suspension) from 6 to 12 months
  Arms: infant placebo
Behavioral: exclusive breastfeeding until 6 months of age — Breastfeeding for 6 months, followed by formula feeding for 6 month. Breastfeeding infants will be prophylaxed with maternal highly active antiretroviral therapy (HAART) (if available) or with infant nevirapine.
  Arms: exclusive breastfeeding for 6 months
Behavioral: breastfeeding for 12 months — Breastfeeding infants will be prophylaxed with maternal HAART (if available) or with infant nevirapine.
  Arms: exclusive breastfeeding for 12 months

SUMMARY:
The purpose of this study is to find ways to improve infant health and survival among infants whose mothers are HIV-infected but who do not themselves have HIV.

DETAILED DESCRIPTION:
As improved MTCT prevention interventions reduce the number of HIV-infected infants in the antepartum and peripartum periods, interventions to improve HIV-free survival among HIV-uninfected infants are needed. Morbidity and mortality are increased among HIV-uninfected infants born to HIV-infected mothers, and reduced infant survival among HIV-exposed infants may lead to as many deaths as HIV infection itself. In Botswana, the use of formula feeding or shorter breastfeeding may worsen the problem of early infant mortality among HIV-exposed infants.

The study will enroll pregnant or postpartum HIV-1-infected women, and their HIV-uninfected infants in Botswana. At 2-4 weeks of age, live HIV-uninfected infants will be randomized to receive either double-blinded cotrimoxazole (CTX) or placebo from 2-4 weeks through 15 months. In addition, breastfeeding (BF) infants will be randomized to BF until either 6 or 12 months of age. Children will be followed prospectively until 18 months of age. The primary endpoint will be survival at 18 months comparing all infants in the CTX vs. placebo arms, and by randomized duration of BF among those BF at randomization. Secondary endpoints will evaluate survival and morbidity/mortality at 12 and 15 months; HIV-free survival to 18 months; and the safety of CTX prophylaxis. Secondary observational objectives include comparing MTCT and mortality by initial feeding method (formula feeding or any BF > 1 month), and an analysis of maternal characteristics as predictors for initial feeding choice and HIV-free survival. All women and infants will receive standard antenatal and peripartum prophylaxis from the Botswana government for MTCT prevention (PMTCT), and will choose a feeding method with counseling. Breastfeeding infants will receive infant nevirapine (NVP) prophylaxis or will be protected from MTCT by the use of maternal HAART.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected women, > 26 weeks gestation and < 34 days postpartum.
* Women must be ¬> 18 years of age and willing/able to sign informed consent.
* Women and infants must be able to follow up regularly at a study clinic through 18 months postpartum.
* For Feeding Randomization Only: Women must be willing to breastfeed for up to 12 months, and to stop at 6 months, depending upon their feeding assignment.

Exclusion Criteria:

* Antepartum women: Known infant anomalies resulting in a high probability that the infant will not survive to 18 months.
* Postpartum women: Known HIV-infected infant, or infant medical condition making survival to 18 months unlikely.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3724 (Estimated)
Dates: Start 2011-05; Primary Completion 2015-03 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Survival | 18 months of age
  The primary outcome measure is survival at 18 months comparing all infants in the CTX vs. placebo arms, and by randomized duration of breastfeeding among those breastfeeding at randomization.

SECONDARY OUTCOMES:
HIV-free Survival | 18 months of age
  Secondary outcome measures will evaluate HIV-free survival between 4 weeks and 18 months among infants randomized to either 6 months or 12 months of breastfeeding.
Safety of CTX prophylaxis | 18 months
  Secondary outcome measures will evaluate the safety of CTX prophylaxis through 18 months
Morbidity and mortality | 18 months of age
  Secondary outcome measures will evaluate morbidity and mortality to 18 months.

CONTACTS AND LOCATIONS:
Overall Officials: Shahin Lockman, MD, MS, Principal Investigator — Harvard School of Public Health (HSPH); Roger L Shapiro, MD, MPH, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (3):
- Botswana (3):
  - Princess Marina Hospital, Gaborone
  - Athlone Hospital, Lobatse
  - Scottish Livingstone Hospital, Molepolole

REFERENCES:
- [Derived] Powis KM, Souda S, Lockman S, Ajibola G, Bennett K, Leidner J, Hughes MD, Moyo S, van Widenfelt E, Jibril HB, Makhema J, Essex M, Shapiro RL. Cotrimoxazole prophylaxis was associated with enteric commensal bacterial resistance among HIV-exposed infants in a randomized controlled trial, Botswana. J Int AIDS Soc. 2017 Nov;20(3):e25021. doi: 10.1002/jia2.25021. PMID 29119726
- [Derived] Lockman S, Hughes M, Powis K, Ajibola G, Bennett K, Moyo S, van Widenfelt E, Leidner J, McIntosh K, Mazhani L, Makhema J, Essex M, Shapiro R. Effect of co-trimoxazole on mortality in HIV-exposed but uninfected children in Botswana (the Mpepu Study): a double-blind, randomised, placebo-controlled trial. Lancet Glob Health. 2017 May;5(5):e491-e500. doi: 10.1016/S2214-109X(17)30143-2. PMID 28395844
- [Derived] Ajibola G, Zash R, Shapiro RL, Batlang O, Botebele K, Bennett K, Chilisa F, Widenfelt EV, Makhema J, Lockman S, Holmes LB, Powis KM. Detecting congenital malformations - Lessons learned from the Mpepu study, Botswana. PLoS One. 2017 Mar 24;12(3):e0173800. doi: 10.1371/journal.pone.0173800. eCollection 2017. PMID 28339500
- See also: Shapiro RL et al. Similar mortality with cotrimoxazole vs. placebo in HIV-exposed uninfected children, Conference on Retroviruses and Opportunistic Infections (CROI 2016), Boston, abstract 37. — http://www.croiconference.org/sessions/similar-mortality-cotrimoxazole-vs-placebo-hiv-exposed-uninfected-children

DOCUMENTS (1):
  • Informed Consent Form (2013-05-22): https://cdn.clinicaltrials.gov/large-docs/61/NCT01229761/ICF_000.pdf